CLINICAL TRIAL: NCT01104558
Title: Association Between Beta-1 and Beta-2 Adrenergic Receptor Polymorphism and Beta-blocker (Bisoprolol) Therapy in Heart Failure
Brief Title: Association Between Genetic Polymorphism of Beta-adrenergic Receptor and Effects of Bisoprolol in Korean Heart Failure Patients.
Acronym: ABBA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMD084000-500
Record Dates: First submitted 2010-02-24; First posted 2010-04-15 (Estimated); Results first posted 2012-04-10 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Heart Failure
Keywords: Bisoprolol; Chronic Heart failure
MeSH Terms: interventions — Bisoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Bisoprolol — Bisoprolol will be given in a starting dose of 1.25 milligram (mg) once daily for two weeks and if it is well tolerated, the dose will be increased to 2.5 mg, 3.75 mg, 5 mg once daily in intervals of two weeks, 5 mg daily as a maintenance therapy. If the subject is tolerable, the dose can be increased as 10 mg/day as maximum dose.
  Other Names: Concor

SUMMARY:
At present, there is some clinical data for different functional response to beta-blockers associated with beta-adrenergic receptor polymorphisms. But there has been no data reported, about the incidence of beta-adrenergic receptor polymorphism and association with beta-adrenergic receptor polymorphism and response to beta-blocker therapy in Korean heart failure (HF) subjects. This single-arm, open-label, multicentric study is designed with the purpose of analyzing the association between genetic polymorphism of beta-adrenergic receptor and the effects of beta-blocker (bisoprolol) in Korean HF subjects.

DETAILED DESCRIPTION:
Heart failure impairs the quality of life of an individual and is considered to be the main cause of morbidity and mortality. Prognosis of HF subjects depends on severity, age and sex. Subjects with HF require lifelong treatment. Pharmacological treatment aims to improve both the quality of life and survival of HF subjects.

OBJECTIVES:

Primary objective:

* To analyze the association between genetic polymorphism of beta-adrenergic receptor and the effects of beta-blocker (bisoprolol) in Korean HF subjects

Secondary objective:

* The frequency of polymorphism of beta adrenergic receptor in Korean HF subjects
* To evaluate change from baseline in 6-minute walking test, heart rate (HR), blood pressure (BP), pro B-type natriuretic peptide (BNP) level at week 26 or End of Treatment (EOT)
* To compare frequency and duration of hospitalization due to heart failure

The method involved in this study will be as follows:

* Initial evaluation of HF subjects
* Blood genomic deoxyribonucleic acid (DNA) isolation and collection
* Bisoprolol treatment as add on therapy with standard treatment for HF subject for 6 months
* Genotype of beta adrenergic receptor polymorphism
* Follow up evaluation of treated subjects

Bisoprolol will be given in a starting dose of 1.25 milligram (mg) once daily for two weeks and if it is well tolerated, the dose will be increased to 2.5 mg, 3.75 mg, 5 mg once daily in intervals of two weeks, 5 mg daily as a maintenance therapy. If the subject is tolerable, the dose can be increased as 10 mg/day as maximum dose.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age and <80 years of age
* Chronic heart failure subjects with stable clinical condition
* New York Heart Association (NYHA) functional classification II-III
* Left ventricular ejection fraction (LVEF) ≤45%

Exclusion Criteria:

* NYHA functional classification IV
* Acute myocardial infarction, Unstable Angina Pectoris, Coronary artery bypass graft, Percutaneous coronary intervention (PCI), Valve surgery in the preceding 3 months
* Hypersensitivity to bisoprolol or any of the Concor excipients
* Subjects with over mild valvular stenosis and severe(Grade III/IV) pulmonary insufficiency
* Systolic Blood Pressure <90 millimeters of mercury (mmHg) at screening
* Resting Heart Rate <55 beats per minute (bpm) confirmed by electrocardiogram (ECG) at screening
* Subjects who are taking concomitant drug which can have drug-drug interaction (DDI) with bisoprolol
* Woman of childbearing age without effective contraception measures, or who are pregnant or lactating

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Ltd.
Locations (1):
- The Catholic University of Korea Seoul St. Mary's Hospital, 505, Banpodong, SeoChoGu, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 117 participants were screened for the study, out of which 17 were screen failures and 100 participants received the study medication.
Groups:
- Bisoprolol: Bisoprolol tablet administered at a starting dose of 1.25 milligram (mg) once daily (OD) for two weeks and if it was well tolerated, the dose was increased to 2.5 mg , 3.75 mg, 5 mg OD in intervals of two weeks, 5 mg OD as a maintenance therapy, for a total time period of 26 weeks. If it was well tolerated, the dose was increased to a maximum of 10 mg/day.
Period: Overall Study
Arm/Group | Bisoprolol
Started | 100
Completed | 83
Not Completed | 17
Not completed — Protocol Violation | 6
Not completed — Missing of primary efficacy assessment | 10
Not completed — Missing of genetic analysis results | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bisoprolol
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.05 (13.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 71

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Echocardiographic Left Ventricular Ejection Fraction (LVEF) According to the Genetic Polymorphism of Beta-1 Adrenergic Receptor-CG at Week 26 or End of Treatment (EOT)
Time Frame: Baseline and Week 26 (or EOT)
Population: Efficacy intention to treat (ITT) population: all enrolled participants; treated with study drug; did not violate inclusion/exclusion criteria; and received primary efficacy assessment at least once after administration. "n" signifies number of participants with particular genotype and were evaluated for this outcome at particular time point.
Measure: Mean (Standard Deviation); unit: Percent LVEF
Arm/Group | Bisoprolol
Number analyzed (Participants) | 83
Percent LVEF
  Baseline: Arg389Arg (n= 53) | 32.44 (7.84)
  Baseline: Arg389Gly (n= 25) | 32.89 (7.70)
  Baseline: Gly389Gly (n= 5) | 32.20 (6.83)
  Change at Week 26 or EOT: Arg389Arg (n= 53) | -8.44 (9.00)
  Change at Week 26 or EOT: Arg389Gly (n= 25) | -9.36 (7.62)
  Change at Week 26 or EOT: Gly389Gly (n= 5) | -9.20 (5.63)

2. Secondary Outcome: Number of Participants With Hospitalization Due to Heart Failure
Time Frame: Baseline to Week 26 (or EOT)
Population: Efficacy ITT population: all enrolled participants; treated with study drug; did not violate inclusion/exclusion criteria; and received primary efficacy assessment at least once after administration.
Measure: Number; unit: Participants
Arm/Group | Bisoprolol
Number analyzed (Participants) | 83
Participants | 1

3. Secondary Outcome: Duration of Hospitalization Due to Heart Failure
Time Frame: Baseline to Week 26 (or EOT)
Population: Participant analyzed included 1 participant from the efficacy ITT population who was hospitalized once due to heart failure.
Measure: Number; unit: Days
Arm/Group | Bisoprolol
Number analyzed (Participants) | 1
Days | 41

4. Secondary Outcome: Change From Baseline in 6-minute Walking Test (6-MWT) Distance According to the Genetic Polymorphism of Beta-1 Adrenergic Receptor-CG at Week 26 or EOT
Description: 6 MWT distance was the distance that a participant could walk in 6 minutes. Participants were asked to perform the test at a pace that was comfortable to them, with as many breaks as they needed.
Time Frame: Baseline and Week 26 (or EOT)
Population: Efficacy ITT population. N (number of participants analyzed) signifies those participants who were evaluated for this measure. "n" signifies number of participants with particular genotype and were evaluated for this outcome at particular time point.
Measure: Mean (Standard Deviation); unit: Meter
Arm/Group | Bisoprolol
Number analyzed (Participants) | 82
Meter
  Baseline: Arg389Arg (n= 53) | 401.36 (161.88)
  Baseline: Arg389Gly (n= 24) | 381.71 (172.47)
  Baseline: Gly389Gly (n= 5) | 371.70 (128.16)
  Change at Week 26 or EOT: Arg389Arg (n= 53) | -20.85 (89.52)
  Change at Week 26 or EOT: Arg389Gly (n= 24) | -0.90 (93.04)
  Change at Week 26 or EOT: Gly389Gly (n= 5) | -20.10 (27.35)

5. Secondary Outcome: Change From Baseline in 6-MWT Distance According to the Genetic Polymorphism of Beta-2 Adrenergic Receptor-AG at Week 26 or EOT
Description: as for outcome 4
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Meter
Arm/Group | Bisoprolol
Number analyzed (Participants) | 82
Meter
  Baseline: Arg16Arg (n= 14) | 449.43 (109.90)
  Baseline: Arg16Gly (n= 41) | 414.73 (155.27)
  Baseline: Gly16Gly (n= 27) | 333.19 (179.71)
  Change at Week 26 or EOT: Arg16Arg (n= 14) | 0.46 (56.91)
  Change at Week 26 or EOT: Arg16Gly (n= 41) | -12.18 (73.57)
  Change at Week 26 or EOT: Gly16Gly (n= 27) | -27.20 (117.54)

6. Primary Outcome: Change From Baseline in Echocardiographic LVEF According to the Genetic Polymorphism of Beta-2 Adrenergic Receptor-AG at Week 26 or EOT
Time Frame: Baseline and Week 26 (or EOT)
Population: Efficacy ITT population: all enrolled participants; treated with study drug; did not violate inclusion/exclusion criteria; and received primary efficacy assessment at least once after administration. "n" signifies number of participants with particular genotype and were evaluated for this outcome at particular time point.
Measure: Mean (Standard Deviation); unit: Percent LVEF
Arm/Group | Bisoprolol
Number analyzed (Participants) | 83
Percent LVEF
  Baseline: Arg16Arg (n= 14) | 31.31 (8.97)
  Baseline: Arg16Gly (n= 41) | 32.67 (7.55)
  Baseline: Gly16Gly (n= 28) | 33.03 (7.35)
  Change at Week 26 or EOT: Arg16Arg (n= 14) | -9.39 (8.49)
  Change at Week 26 or EOT: Arg16Gly (n= 41) | -7.87 (8.94)
  Change at Week 26 or EOT: Gly16Gly (n= 28) | -9.76 (7.57)

7. Primary Outcome: Change From Baseline in Echocardiographic LVEF According to the Genetic Polymorphism of Beta-2 Adrenergic Receptor-CG at Week 26 or EOT
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percent LVEF
Arm/Group | Bisoprolol
Number analyzed (Participants) | 83
Percent LVEF
  Baseline: Glu27Glu (n= 1) | 38.00 (NA) — The standard deviation was not available because there was only 1 participant with this particular genotype.
  Baseline: Glu27Gln (n= 15) | 33.01 (7.30)
  Baseline: Gln27Gln (n= 67) | 32.38 (7.82)
  Change at Week 26 or EOT: Glu27Glu (n= 1) | -13.00 (NA) — The standard deviation was not available because there was only 1 participant with this particular genotype.
  Change at Week 26 or EOT: Glu27Gln (n= 15) | -8.71 (5.73)
  Change at Week 26 or EOT: Gln27Gln (n= 67) | -8.71 (8.94)

8. Primary Outcome: Change From Baseline in Echocardiographic LVEF According to the Genetic Polymorphism of G Protein-coupled Receptor Kinase 5 (GRK5)-AG at Week 26 or EOT
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percent LVEF
Arm/Group | Bisoprolol
Number analyzed (Participants) | 83
Percent LVEF
  Baseline: GRK5-Arg304 (n= 50) | 32.37 (7.81)
  Baseline: GRK5-Arg304His (n= 30) | 33.14 (7.46)
  Baseline: GRK5-His304 (n= 3) | 29.87 (9.33)
  Change at Week 26 or EOT: GRK5-Arg304 (n= 50) | -7.69 (7.73)
  Change at Week 26 or EOT: GRK5-Arg304His (n= 30) | -10.19 (8.93)
  Change at Week 26 or EOT: GRK5-His304 (n= 3) | -12.47 (13.27)

9. Secondary Outcome: Change From Baseline in 6-MWT Distance According to the Genetic Polymorphism of Beta-2 Adrenergic Receptor-CG at Week 26 or EOT
Description: as for outcome 4
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Meter
Arm/Group | Bisoprolol
Number analyzed (Participants) | 82
Meter
  Baseline: Glu27Glu (n= 1) | 468.00 (NA) — The standard deviation was not available because there was only 1 participant with this particular genotype.
  Baseline: Glu27Gln (n= 15) | 404.63 (175.65)
  Baseline: Gln27Gln (n= 66) | 390.22 (160.83)
  Change at Week 26 or EOT: Glu27Glu (n= 1) | -57.00 (NA) — The standard deviation was not available because there was only 1 participant with this particular genotype.
  Change at Week 26 or EOT: Glu27Gln (n= 15) | 12.23 (106.68)
  Change at Week 26 or EOT: Gln27Gln (n= 66) | -20.51 (83.33)

10. Secondary Outcome: Change From Baseline in 6-minute Walking Test (6-MWT) Distance According to the Genetic Polymorphism of GRK5-AG at Week 26 or EOT
Description: as for outcome 4
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Meter
Arm/Group | Bisoprolol
Number analyzed (Participants) | 82
Meter
  Baseline: GRK5-Arg304 (n= 49) | 390.68 (160.61)
  Baseline: GRK5-Arg304His (n= 30) | 395.11 (173.68)
  Baseline: GRK5-His304 (n= 3) | 431.67 (42.52)
  Change at Week 26 or EOT: GRK5-Arg304 (n= 49) | -13.86 (79.64)
  Change at Week 26 or EOT: GRK5-Arg304His (n= 30) | -17.61 (104.93)
  Change at Week 26 or EOT: GRK5-His304 (n= 3) | -6.67 (25.66)

11. Secondary Outcome: Change From Baseline in Heart Rate (6 MWT- Before Walking) According to the Genetic Polymorphism of Beta-1 Adrenergic Receptor-CG at Week 26 or EOT
Description: The change in heart rate was calculated as 6-MWT before walking heart rate at Week 26 minus 6-MWT before walking heart rate at baseline.
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | Bisoprolol
Number analyzed (Participants) | 82
Beats per minute (bpm)
  Baseline: Arg389Arg (n= 53) | 76.47 (12.90)
  Baseline: Arg389Gly (n= 24) | 82.25 (14.66)
  Baseline: Gly389Gly (n= 5) | 83.20 (19.52)
  Change at Week 26 or EOT: Arg389Arg (n= 53) | 8.91 (14.80)
  Change at Week 26 or EOT: Arg389Gly (n= 24) | 11.79 (15.13)
  Change at Week 26 or EOT: Gly389Gly (n= 5) | 12.00 (22.55)

12. Secondary Outcome: Change From Baseline in Heart Rate (6 MWT- Before Walking) According to the Genetic Polymorphism of Beta-2 Adrenergic Receptor-AG at Week 26 or EOT
Description: as for outcome 11
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Bisoprolol
Number analyzed (Participants) | 82
bpm
  Baseline: Arg16Arg (n= 14) | 79.21 (13.96)
  Baseline: Arg16Gly (n= 41) | 79.02 (15.06)
  Baseline: Gly16Gly (n= 27) | 77.56 (12.61)
  Change at Week 26 or EOT: Arg16Arg (n= 14) | 13.21 (12.71)
  Change at Week 26 or EOT: Arg16Gly (n= 41) | 9.20 (13.88)
  Change at Week 26 or EOT: Gly16Gly (n= 27) | 9.37 (18.45)

13. Secondary Outcome: Change From Baseline in Heart Rate (6 MWT- Before Walking) According to the Genetic Polymorphism of Beta-2 Adrenergic Receptor-CG at Week 26 or EOT
Description: as for outcome 11
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Bisoprolol
Number analyzed (Participants) | 82
bpm
  Baseline: Glu27Glu (n= 1) | 92.00 (NA) — The standard deviation was not available because there was only 1 participant with this particular genotype.
  Baseline: Glu27Gln (n= 15) | 76.60 (11.47)
  Baseline: Gln27Gln (n= 66) | 78.82 (14.52)
  Change at Week 26 or EOT: Glu27Glu (n= 1) | 9.00 (NA) — The standard deviation was not available because there was only 1 participant with this particular genotype.
  Change at Week 26 or EOT: Glu27Gln (n= 15) | 10.33 (15.77)
  Change at Week 26 or EOT: Gln27Gln (n= 66) | 9.86 (15.37)

14. Secondary Outcome: Change From Baseline in Heart Rate (6 MWT- Before Walking) According to the Genetic Polymorphism of GRK5-AG at Week 26 or EOT
Description: as for outcome 11
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Bisoprolol
Number analyzed (Participants) | 82
bpm
  Baseline: GRK5-Arg304 (n= 49) | 77.29 (12.29)
  Baseline: GRK5-Arg304His (n= 30) | 80.80 (16.54)
  Baseline: GRK5-His304 (n= 3) | 77.33 (13.32)
  Change at Week 26 or EOT: GRK5-Arg304 (n= 49) | 10.92 (13.00)
  Change at Week 26 or EOT: GRK5-Arg304His (n= 30) | 7.83 (18.69)
  Change at Week 26 or EOT: GRK5-His304 (n= 3) | 15.00 (13.00)

15. Secondary Outcome: Change From Baseline in Heart Rate (6 MWT- After Walking) According to the Genetic Polymorphism of Beta-1 Adrenergic Receptor-CG at Week 26 or EOT
Description: The change in heart rate was calculated as 6-MWT after walking heart rate at Week 26 minus 6-MWT after walking heart rate at baseline.
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Bisoprolol
Number analyzed (Participants) | 82
bpm
  Baseline: Arg389Arg (n= 53) | 92.02 (19.82)
  Baseline: Arg389Gly (n= 24) | 90.92 (21.37)
  Baseline: Gly389Gly (n= 5) | 92.80 (25.99)
  Change at Week 26 or EOT: Arg389Arg (n= 53) | 11.83 (17.83)
  Change at Week 26 or EOT: Arg389Gly (n= 24) | 15.88 (16.54)
  Change at Week 26 or EOT: Gly389Gly (n= 5) | 4.60 (15.79)

16. Secondary Outcome: Change From Baseline in Heart Rate (6 MWT- After Walking) According to the Genetic Polymorphism of Beta-2 Adrenergic Receptor-AG at Week 26 or EOT
Description: as for outcome 15
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Bisoprolol
Number analyzed (Participants) | 82
bpm
  Baseline: Arg16Arg (n= 14) | 87.86 (18.53)
  Baseline: Arg16Gly (n= 41) | 95.05 (21.41)
  Baseline: Gly16Gly (n= 27) | 88.74 (19.55)
  Change at Week 26 or EOT: Arg16Arg (n= 14) | 11.21 (15.34)
  Change at Week 26 or EOT: Arg16Gly (n= 41) | 12.37 (18.83)
  Change at Week 26 or EOT: Gly16Gly (n= 27) | 13.59 (16.57)

17. Secondary Outcome: Change From Baseline in Heart Rate (6 MWT- After Walking) According to the Genetic Polymorphism of Beta-2 Adrenergic Receptor-CG at Week 26 or EOT
Description: as for outcome 15
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Bisoprolol
Number analyzed (Participants) | 82
bpm
  Baseline: Glu27Glu (n= 1) | 90.00 (NA) — The standard deviation was not available because there was only 1 participant with this particular genotype.
  Baseline: Glu27Gln (n= 15) | 84.40 (15.89)
  Baseline: Gln27Gln (n= 66) | 93.44 (21.16)
  Change at Week 26 or EOT: Glu27Glu (n= 1) | -3.00 (NA) — The standard deviation was not available because there was only 1 participant with this particular genotype.
  Change at Week 26 or EOT: Glu27Gln (n= 15) | 9.73 (13.10)
  Change at Week 26 or EOT: Gln27Gln (n= 66) | 13.45 (18.24)

18. Secondary Outcome: Change From Baseline in Heart Rate (6 MWT- After Walking) According to the Genetic Polymorphism of GRK5-AG at Week 26 or EOT
Description: as for outcome 15
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Bisoprolol
Number analyzed (Participants) | 82
bpm
  Baseline: GRK5-Arg304 (n= 49) | 92.41 (20.87)
  Baseline: GRK5-Arg304His (n= 30) | 89.30 (19.18)
  Baseline: GRK5-His304 (n= 3) | 105.33 (25.70)
  Change at Week 26 or EOT: GRK5-Arg304 (n= 49) | 14.59 (16.16)
  Change at Week 26 or EOT: GRK5-Arg304His (n= 30) | 8.53 (19.39)
  Change at Week 26 or EOT: GRK5-His304 (n= 3) | 20.00 (8.54)

19. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) (6 MWT- Before Walking) According to the Genetic Polymorphism of Beta-1 Adrenergic Receptor-CG at Week 26 or EOT
Description: The change in SBP was calculated as 6-MWT before walking SBP at Week 26 minus 6-MWT before walking SBP at baseline.
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Bisoprolol
Number analyzed (Participants) | 81
millimeters of mercury (mmHg)
  Baseline: Arg389Arg (n= 52) | 121.81 (19.07)
  Baseline: Arg389Gly (n= 24) | 123.54 (15.91)
  Baseline: Gly389Gly (n= 5) | 117.40 (15.09)
  Change at Week 26 or EOT: Arg389Arg (n= 52) | -0.96 (15.09)
  Change at Week 26 or EOT: Arg389Gly (n= 24) | -2.75 (16.54)
  Change at Week 26 or EOT: Gly389Gly (n= 5) | -0.40 (25.07)

20. Secondary Outcome: Change From Baseline in SBP (6 MWT- Before Walking) According to the Genetic Polymorphism of Beta-2 Adrenergic Receptor-AG at Week 26 or EOT
Description: The change in SBP was calculated as 6-MWT before walking SBP at Week 26 minus 6-MWT before walking SBP at baseline.
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol
Number analyzed (Participants) | 81
mmHg
  Baseline: Arg16Arg (n= 14) | 132.36 (27.18)
  Baseline: Arg16Gly (n= 41) | 117.83 (14.61)
  Baseline: Gly16Gly (n= 26) | 123.15 (14.22)
  Change at Week 26 or EOT: Arg16Arg (n= 14) | 2.50 (15.62)
  Change at Week 26 or EOT: Arg16Gly (n= 41) | -4.32 (15.69)
  Change at Week 26 or EOT: Gly16Gly (n= 26) | 0.92 (16.43)

21. Secondary Outcome: Change From Baseline in SBP (6 MWT- Before Walking) According to the Genetic Polymorphism of Beta-2 Adrenergic Receptor-CG at Week 26 or EOT
Description: The change in SBP was calculated as 6-MWT before walking SBP at Week 26 minus 6-MWT before walking SBP at baseline.
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol
Number analyzed (Participants) | 81
mmHg
  Baseline: Glu27Glu (n= 1) | 130.00 (NA) — The standard deviation was not available because there was only 1 participant with this particular genotype.
  Baseline: Glu27Gln (n= 15) | 115.53 (11.55)
  Baseline: Gln27Gln (n= 65) | 123.43 (18.85)
  Change at Week 26 or EOT: Glu27Glu (n= 1) | -13.00 (NA) — The standard deviation was not available because there was only 1 participant with this particular genotype.
  Change at Week 26 or EOT: Glu27Gln (n= 15) | -4.33 (12.31)
  Change at Week 26 or EOT: Gln27Gln (n= 65) | -0.62 (16.79)

22. Secondary Outcome: Change From Baseline in SBP (6 MWT- Before Walking) According to the Genetic Polymorphism of GRK5-AG at Week 26 or EOT
Description: The change in SBP was calculated as 6-MWT before walking SBP at Week 26 minus 6-MWT before walking SBP at baseline.
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol
Number analyzed (Participants) | 81
mmHg
  Baseline: GRK5-Arg304 (n= 48) | 118.92 (13.79)
  Baseline: GRK5-Arg304His (n= 30) | 126.53 (22.61)
  Baseline: GRK5-His304 (n= 3) | 127.33 (16.17)
  Change at Week 26 or EOT: GRK5-Arg304 (n= 48) | -2.25 (15.86)
  Change at Week 26 or EOT: GRK5-Arg304His (n= 30) | -1.13 (16.78)
  Change at Week 26 or EOT: GRK5-His304 (n= 3) | 8.00 (9.64)

23. Secondary Outcome: Change From Baseline in SBP (6 MWT- After Walking) According to the Genetic Polymorphism of Beta-1 Adrenergic Receptor-CG at Week 26 or EOT
Description: The change in SBP was calculated as 6-MWT after walking SBP at Week 26 minus 6-MWT after walking SBP at baseline.
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol
Number analyzed (Participants) | 81
mmHg
  Baseline: Arg389Arg (n= 52) | 128.77 (20.95)
  Baseline: Arg389Gly (n= 24) | 130.25 (22.55)
  Baseline: Gly389Gly (n= 5) | 128.60 (14.52)
  Change at Week 26 or EOT: Arg389Arg (n= 52) | -2.92 (18.24)
  Change at Week 26 or EOT: Arg389Gly (n= 24) | -0.46 (22.31)
  Change at Week 26 or EOT: Gly389Gly (n= 5) | 5.40 (23.64)

24. Secondary Outcome: Change From Baseline in SBP (6 MWT- After Walking) According to the Genetic Polymorphism of Beta-2 Adrenergic Receptor-AG at Week 26 or EOT
Description: The change in SBP was calculated as 6-MWT after walking SBP at Week 26 minus 6-MWT after walking SBP at baseline.
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol
Number analyzed (Participants) | 81
mmHg
  Baseline: Arg16Arg (n= 14) | 138.71 (25.63)
  Baseline: Arg16Gly (n= 41) | 126.56 (19.78)
  Baseline: Gly16Gly (n= 26) | 128.23 (19.19)
  Change at Week 26 or EOT: Arg16Arg (n= 14) | 3.29 (17.79)
  Change at Week 26 or EOT: Arg16Gly (n= 41) | -4.34 (20.96)
  Change at Week 26 or EOT: Gly16Gly (n= 26) | -0.15 (18.59)

25. Secondary Outcome: Change From Baseline in SBP (6 MWT- After Walking) According to the Genetic Polymorphism of Beta-2 Adrenergic Receptor-CG at Week 26 or EOT
Description: The change in SBP was calculated as 6-MWT after walking SBP at Week 26 minus 6-MWT after walking SBP at baseline.
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol
Number analyzed (Participants) | 81
mmHg
  Baseline: Glu27Glu (n= 1) | 113.00 (NA) — The standard deviation was not available because there was only 1 participant with this particular genotype.
  Baseline: Glu27Gln (n= 15) | 124.47 (9.62)
  Baseline: Gln27Gln (n= 65) | 130.54 (22.69)
  Change at Week 26 or EOT: Glu27Glu (n= 1) | -18.00 (NA) — The standard deviation was not available because there was only 1 participant with this particular genotype.
  Change at Week 26 or EOT: Glu27Gln (n= 15) | -4.93 (12.61)
  Change at Week 26 or EOT: Gln27Gln (n= 65) | -0.68 (21.03)

26. Secondary Outcome: Change From Baseline in SBP (6 MWT- After Walking) According to the Genetic Polymorphism of GRK5-AG at Week 26 or EOT
Description: The change in SBP was calculated as 6-MWT after walking SBP at Week 26 minus 6-MWT after walking SBP at baseline.
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol
Number analyzed (Participants) | 81
mmHg
  Baseline: GRK5-Arg304 (n= 48) | 127.52 (17.67)
  Baseline: GRK5-Arg304His (n= 30) | 131.27 (25.87)
  Baseline: GRK5-His304 (n= 3) | 135.33 (16.04)
  Change at Week 26 or EOT: GRK5-Arg304 (n= 48) | -2.10 (20.08)
  Change at Week 26 or EOT: GRK5-Arg304His (n= 30) | -2.37 (19.51)
  Change at Week 26 or EOT: GRK5-His304 (n= 3) | 12.00 (15.10)

27. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) (6 MWT- Before Walking) According to the Genetic Polymorphism of Beta-1 Adrenergic Receptor-CG at Week 26 or EOT
Description: The change in DBP was calculated as 6-MWT before walking DBP at Week 26 minus 6-MWT before walking DBP at baseline.
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol
Number analyzed (Participants) | 81
mmHg
  Baseline: Arg389Arg (n= 52) | 75.69 (14.70)
  Baseline: Arg389Gly (n= 24) | 78.17 (12.33)
  Baseline: Gly389Gly (n= 5) | 79.40 (5.55)
  Change at Week 26 or EOT: Arg389Arg (n= 52) | 0.10 (13.13)
  Change at Week 26 or EOT: Arg389Gly (n= 24) | 0.29 (15.16)
  Change at Week 26 or EOT: Gly389Gly (n= 5) | 0.60 (11.70)

28. Secondary Outcome: Change From Baseline in DBP (6 MWT- Before Walking) According to the Genetic Polymorphism of Beta-2 Adrenergic Receptor-AG at Week 26 or EOT
Description: The change in DBP was calculated as 6-MWT before walking DBP at Week 26 minus 6-MWT before walking DBP at baseline.
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol
Number analyzed (Participants) | 81
mmHg
  Baseline: Arg16Arg (n= 14) | 83.14 (22.76)
  Baseline: Arg16Gly (n= 41) | 75.59 (11.11)
  Baseline: Gly16Gly (n= 26) | 74.85 (9.79)
  Change at Week 26 or EOT: Arg16Arg (n= 14) | 4.07 (18.89)
  Change at Week 26 or EOT: Arg16Gly (n= 41) | -0.88 (10.39)
  Change at Week 26 or EOT: Gly16Gly (n= 26) | -0.23 (14.71)

29. Secondary Outcome: Change From Baseline in DBP (6 MWT- Before Walking) According to the Genetic Polymorphism of Beta-2 Adrenergic Receptor-CG at Week 26 or EOT
Description: The change in DBP was calculated as 6-MWT before walking DBP at Week 26 minus 6-MWT before walking DBP at baseline.
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol
Number analyzed (Participants) | 81
mmHg
  Baseline: Glu27Glu (n= 1) | 68.00 (NA) — The standard deviation was not available because there was only 1 participant with this particular genotype.
  Baseline: Glu27Gln (n= 15) | 71.80 (8.90)
  Baseline: Gln27Gln (n= 65) | 77.91 (14.33)
  Change at Week 26 or EOT: Glu27Glu (n= 1) | -28.00 (NA) — The standard deviation was not available because there was only 1 participant with this particular genotype.
  Change at Week 26 or EOT: Glu27Gln (n= 15) | -1.93 (11.22)
  Change at Week 26 or EOT: Gln27Gln (n= 65) | 1.11 (13.66)

30. Secondary Outcome: Change From Baseline in DBP (6 MWT- Before Walking) According to the Genetic Polymorphism of GRK5-AG at Week 26 or EOT
Description: The change in DBP was calculated as 6-MWT before walking DBP at Week 26 minus 6-MWT before walking DBP at baseline.
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol
Number analyzed (Participants) | 81
mmHg
  Baseline: GRK5-Arg304 (n= 48) | 74.90 (10.79)
  Baseline: GRK5-Arg304His (n= 30) | 78.87 (17.43)
  Baseline: GRK5-His304 (n= 3) | 82.67 (7.02)
  Change at Week 26 or EOT: GRK5-Arg304 (n= 48) | 0.06 (12.93)
  Change at Week 26 or EOT: GRK5-Arg304His (n= 30) | -0.13 (15.17)
  Change at Week 26 or EOT: GRK5-His304 (n= 3) | 5.33 (1.15)

31. Secondary Outcome: Change From Baseline in DBP (6 MWT- After Walking) According to the Genetic Polymorphism of Beta-1 Adrenergic Receptor-CG at Week 26 or EOT
Description: The change in DBP was calculated as 6-MWT after walking DBP at Week 26 minus 6-MWT after walking DBP at baseline.
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol
Number analyzed (Participants) | 81
mmHg
  Baseline: Arg389Arg (n= 52) | 80.15 (13.62)
  Baseline: Arg389Gly (n= 24) | 80.50 (12.60)
  Baseline: Gly389Gly (n= 5) | 81.80 (8.50)
  Change at Week 26 or EOT: Arg389Arg (n= 52) | -0.04 (13.66)
  Change at Week 26 or EOT: Arg389Gly (n= 24) | 3.63 (11.86)
  Change at Week 26 or EOT: Gly389Gly (n= 5) | 1.00 (14.04)

32. Secondary Outcome: Change From Baseline in DBP (6 MWT- After Walking) According to the Genetic Polymorphism of Beta-2 Adrenergic Receptor-AG at Week 26 or EOT
Description: The change in DBP was calculated as 6-MWT after walking DBP at Week 26 minus 6-MWT after walking DBP at baseline.
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol
Number analyzed (Participants) | 81
mmHg
  Baseline: Arg16Arg (n= 14) | 86.14 (18.92)
  Baseline: Arg16Gly (n= 41) | 79.66 (11.67)
  Baseline: Gly16Gly (n= 26) | 78.35 (10.44)
  Change at Week 26 or EOT: Arg16Arg (n= 14) | 4.21 (18.73)
  Change at Week 26 or EOT: Arg16Gly (n= 41) | -0.54 (10.51)
  Change at Week 26 or EOT: Gly16Gly (n= 26) | 2.04 (13.44)

33. Secondary Outcome: Change From Baseline in DBP (6 MWT- After Walking) According to the Genetic Polymorphism of Beta-2 Adrenergic Receptor-CG at Week 26 or EOT
Description: The change in DBP was calculated as 6-MWT after walking DBP at Week 26 minus 6-MWT after walking DBP at baseline.
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol
Number analyzed (Participants) | 81
mmHg
  Baseline: Glu27Glu (n= 1) | 65.00 (NA) — The standard deviation was not available because there was only 1 participant with this particular genotype.
  Baseline: Glu27Gln (n= 15) | 77.40 (6.31)
  Baseline: Gln27Gln (n= 65) | 81.28 (13.94)
  Change at Week 26 or EOT: Glu27Glu (n= 1) | -21.00 (NA) — The standard deviation was not available because there was only 1 participant with this particular genotype.
  Change at Week 26 or EOT: Glu27Gln (n= 15) | 0.87 (10.78)
  Change at Week 26 or EOT: Gln27Gln (n= 65) | 1.51 (13.48)

34. Secondary Outcome: Change From Baseline in DBP (6 MWT- After Walking) According to the Genetic Polymorphism of GRK5-AG at Week 26 or EOT
Description: The change in DBP was calculated as 6-MWT after walking DBP at Week 26 minus 6-MWT after walking DBP at baseline.
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol
Number analyzed (Participants) | 81
mmHg
  Baseline: GRK5-Arg304 (n= 48) | 79.10 (11.08)
  Baseline: GRK5-Arg304His (n= 30) | 81.97 (15.98)
  Baseline: GRK5-His304 (n= 3) | 84.33 (4.04)
  Change at Week 26 or EOT: GRK5-Arg304 (n= 48) | 0.79 (13.46)
  Change at Week 26 or EOT: GRK5-Arg304His (n= 30) | 1.27 (13.31)
  Change at Week 26 or EOT: GRK5-His304 (n= 3) | 4.67 (5.51)

35. Secondary Outcome: Change From Baseline in Pro-B-type Natriuretic Peptide (BNP) Levels According to the Genetic Polymorphism of Beta-1 Adrenergic Receptor-CG at Week 26 or EOT
Description: BNP is a substance secreted from the ventricles or lower chambers of the heart in response to changes in pressure that occur when heart failure develops and worsens. The level of BNP in the blood increases when heart failure symptoms worsen, and decreases when the heart failure condition is stable. The BNP level in a person with heart failure is higher than in a person with normal heart function.
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: picograms (pg)/ milliliter (mL)
Arm/Group | Bisoprolol
Number analyzed (Participants) | 83
picograms (pg)/ milliliter (mL)
  Baseline: Arg389Arg (n= 53) | 1484.02 (3258.55)
  Baseline: Arg389Gly (n= 25) | 851.47 (830.19)
  Baseline: Gly389Gly (n= 5) | 1011.30 (558.49)
  Change at Week 26 or EOT: Arg389Arg (n= 53) | 292.10 (2452.11)
  Change at Week 26 or EOT: Arg389Gly (n= 24) | 310.63 (643.97)
  Change at Week 26 or EOT: Gly389Gly (n= 5) | 394.32 (407.89)

36. Secondary Outcome: Change From Baseline in Pro-BNP Levels According to the Genetic Polymorphism of Beta-2 Adrenergic Receptor-AG at Week 26 or EOT
Description: as for outcome 35
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Bisoprolol
Number analyzed (Participants) | 83
pg/mL
  Baseline: Arg16Arg (n= 14) | 2809.30 (5763.28)
  Baseline: Arg16Gly (n= 41) | 823.71 (809.39)
  Baseline: Gly16Gly (n= 28) | 1139.07 (1691.51)
  Change at Week 26 or EOT: Arg16Arg (n= 14) | 1600.88 (4294.99)
  Change at Week 26 or EOT: Arg16Gly (n= 40) | -33.98 (909.74)
  Change at Week 26 or EOT: Gly16Gly (n= 28) | 137.68 (901.46)

37. Secondary Outcome: Change From Baseline in Pro-BNP Levels According to the Genetic Polymorphism of Beta-2 Adrenergic Receptor-CG at Week 26 or EOT
Description: as for outcome 35
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Bisoprolol
Number analyzed (Participants) | 83
pg/mL
  Baseline: Glu27Glu (n= 1) | 120.80 (NA) — The standard deviation was not available because there was only 1 participant with this particular genotype.
  Baseline: Glu27Gln (n= 15) | 878.31 (919.99)
  Baseline: Gln27Gln (n= 67) | 1368.67 (2915.35)
  Change at Week 26 or EOT: Glu27Glu (n= 1) | 84.91 (NA) — The standard deviation was not available because there was only 1 participant with this particular genotype.
  Change at Week 26 or EOT: Glu27Gln (n= 15) | 131.60 (902.50)
  Change at Week 26 or EOT: Gln27Gln (n= 66) | 346.20 (2187.04)

38. Secondary Outcome: Change From Baseline in Pro-BNP Levels According to the Genetic Polymorphism of GRK5-AG at Week 26 or EOT
Description: as for outcome 35
Time Frame: Baseline and Week 26 (or EOT)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Bisoprolol
Number analyzed (Participants) | 83
pg/mL
  Baseline: GRK5-Arg304 (n= 50) | 895.52 (1291.90)
  Baseline: GRK5-Arg304His (n= 30) | 1854.63 (4030.43)
  Baseline: GRK5-His304 (n= 3) | 1527.09 (1836.19)
  Change at Week 26 or EOT: GRK5-Arg304 (n= 49) | -33.78 (850.25)
  Change at Week 26 or EOT: GRK5-Arg304His (n= 30) | 799.31 (3052.03)
  Change at Week 26 or EOT: GRK5-His304 (n= 3) | 861.39 (1450.04)

ADVERSE EVENTS:
Time Frame: Up to Week 26 (or EOT)
Description: An adverse event (AE) was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an Investigational Medicinal Product (IMP), regardless of causal relationship and even if no IMP has been administered.
Arm/Group | Bisoprolol
Serious Adverse Events (participants affected / at risk) | 7/100
Other Adverse Events (participants affected / at risk) | 93/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bisoprolol (N=100)
Death sudden (General disorders) | 1
Edema limbs (General disorders) | 1
INR increased (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Hospitalisation (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bisoprolol (N=100)
Bradycardia (Cardiac disorders) | 2
Chest discomfort (Cardiac disorders) | 6
Chest pain (Cardiac disorders) | 6
Diabetic retinopathy (Eye disorders) | 1
Keratitis (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Epigastric discomfort (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 1
General body pain (General disorders) | 1
Pitting edema (General disorders) | 1
Weakness generalized (General disorders) | 2
Herpes zoster (Infections and infestations) | 2
Liver function test abnormal (Investigations) | 1
Weight increased (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Back discomfort (Musculoskeletal and connective tissue disorders) | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 10
Dysarthria (Nervous system disorders) | 1
Head discomfort (Nervous system disorders) | 1
Near syncope (Nervous system disorders) | 1
Orthostatic dizziness (Nervous system disorders) | 1
Sleepiness (Nervous system disorders) | 1
Slurred speech (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Tingling feet/hands (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 2
Voiding difficulty (Renal and urinary disorders) | 1
Nipple pain (Reproductive system and breast disorders) | 1
Common cold (Respiratory, thoracic and mediastinal disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dry cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Sputum (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other